CLINICAL TRIAL: NCT00807859
Title: An Open-Label Study of AMG 386 in Combination With Either Paclitaxel and Trastuzumab or Capecitabine and Lapatinib in Subjects With HER2-positive Locally Recurrent or Metastatic Breast Cancer
Brief Title: Safety Study of AMG 386 to Treat HER2-positive Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20062042
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Tumors; Cancer; Locally Recurrent and Metastatic Breast Cancer; Metastases; Metastatic Cancer; Oncology; Solid Tumors; Tumors
Keywords: AMG 386; Paclitaxel; Trastuzumab; Capecitabine; Lapatinib; HER2-positive; metastatic breast cancer; locally recurrent breast cancer; Taxol; Herceptin; Xeloda; Tykerb; anti-angiogenic therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — trebananib; Paclitaxel; Trastuzumab; Capecitabine; Lapatinib

ARMS (4):
- Cohort A1 (Experimental)
  Interventions: Drug: AMG 386 10 mgkg, Paclitaxel and Trastuzumab
- Cohort A3 (Experimental)
  Interventions: Drug: AMG 386 30 mg/kg, Paclitaxel and Trastuzumab
- Cohort B1 (Experimental)
  Interventions: Drug: AMG 386 10 mg/kg, Capecitabine and Lapatinib
- Cohort B3 (Experimental)
  Interventions: Drug: AMG 386 30 mg/kg, Capecitabine and Lapatinib

INTERVENTIONS:
Drug: AMG 386 30 mg/kg, Paclitaxel and Trastuzumab — AMG 386 30 mg/kg IV QW, paclitaxel 80 mg/m2 IV QW, trastuzumab: initial dose 8 mg/kg IV week 1, then 6 mg/kg IV Q3W
  Arms: Cohort A3
Drug: AMG 386 30 mg/kg, Capecitabine and Lapatinib — AMG 386 30 mg/kg IV QW, capecitabine 2000 mg/m2 divided into 2 doses given PO Q12 hrs, days 1-14 every 21 days, lapatinib 1250 mg PO QD
  Arms: Cohort B3
Drug: AMG 386 10 mgkg, Paclitaxel and Trastuzumab — AMG 386 10 mg/kg IV QW, paclitaxel 80 mg/m2 IV QW, trastuzumab: initial dose 8 mg/kg IV week 1, then 6 mg/kg IV Q3W
  Arms: Cohort A1
Drug: AMG 386 10 mg/kg, Capecitabine and Lapatinib — AMG 386 10 mg/kg IV QW, capecitabine 2000 mg/m2 divided into 2 doses given PO Q12 hrs, days 1-14 every 21 days, lapatinib 1250 mg PO QD
  Arms: Cohort B1

SUMMARY:
The purpose of this study is to determine if AMG 386 in combination with either paclitaxel and trastuzumab or capecitabine and lapatinib is safe and well tolerated in subjects with HER2-positive locally recurrent or metastatic breast cancer.

This is an open-label phase 1b trial and has 2 study parts. Study part 1 is a dose escalation study to determine a tolerable dose of AMG 386 in combination with paclitaxel and trastuzumab (cohort A) or with capecitabine and lapatinib (cohort B). Study part 2 is cohort expansion of the tolerable doses determined in part 1.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease not amenable to any local treatment with curative intent.
* HER2-positive by FISH, CISH, or IHC 3+
* ECOG performance status 0 or 1
* Left ventricular ejection fraction greater than or equal to institutional lower limit of normal
* Adequate laboratory studies (hematological, chemistries and urinalysis)
* Life expectancy greater than or equal to 3 months
* Cohort A only:
* Trastuzumab naïve or trastuzumab in the neo-adjuvant setting
* No clinically significant drop in cardiac function prior exposure to trastuzumab
* No prior chemotherapy for metastatic or locally recurrent breast cancer
* No prior lapatinib therapy
* At least 3 weeks from enrollment since prior chemotherapeutic agents, including taxanes, in the neoadjuvant or adjuvant setting
* At least 3 months from enrollment since prior trastuzumab in the neoadjuvant or adjuvant setting
* Cohort B only:
* Must have failed trastuzumab in the first-line metastatic setting. Trastuzumab must be discontinued for at least 3 weeks prior to enrollment
* Must have received prior chemotherapy as adjuvant therapy or for metastatic disease
* Prior chemotherapy treatment must be discontinued for at least 3 weeks prior to enrollment
* No prior capecitabine
* No prior lapatinib

Exclusion Criteria:

* Inflammatory breast cancer
* Central nervous system metastasis
* Clinically significant cardiovascular disease
* Radiation therapy ≤ 14 days prior to enrollment.
* Concurrent anticoagulation therapy, excluding aspirin, anti-platelet agents, low molecular weight heparin or low dose warfarin per protocol.
* Uncontrolled hypertension defined as diastolic blood pressure > 90 mmHg OR systolic blood pressure > 140 mmHg.
* Subjects with a history of prior malignancy, except:
* For Cohort B only:
* Current or prior history of long QT syndrome
* Baseline ECG report of QTc interval of > 480 milliseconds
* Severe chronic liver disease (Child Pugh C)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03-09 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2015-10-19 (Actual)

PRIMARY OUTCOMES:
Primary objective is to identify the incidence of adverse events and clinical laboratory abnormalities defined as a dose limiting toxicity in subjects treated with AMG 386 plus paclitaxel and trastuzumab or with AMG 386 plus capecitabine and lapatinib | 24 months

SECONDARY OUTCOMES:
To evaluate the incidence of adverse events and clinical laboratory abnormalities not defined as DLTs | 24 months
To evaluate the pharmacokinetics (PK) of AMG 386, trastuzumab, and paclitaxel (cohort A) or AMG 386, lapatinib, and capecitabine (and its active metabolite, 5-FU; cohort B) when administered in combination | 24 months
To estimate the incidence of anti AMG 386 antibody formation | 24 months
To evaluate the treatment effect as measured by the following: objective response rate (ORR), duration of response (DOR), change in tumor burden and progression-free survival (PFS) | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (12):
  - Research Site, Tucson, Arizona
  - Research Site, Boca Raton, Florida
  - Research Site, Iowa City, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Lebanon, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, New City, New York
  - Research Site, New York, New York
  - Research Site, Nyack, New York
  - Research Site, Middletown, Ohio
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Wilrijk
- France (7):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, La Roche-sur-Yon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Pierre BÃ©nite Cedex
  - Research Site, Toulouse

REFERENCES:
- [Background] Kaufman PA, Wildiers H, Freyer G, Kemeny M, Goncalves A, Jerusalem G, Stopeck A, Vrindavanam N, Dalenc F, Nanayakkara N, Wu B, Pickett CA. Phase 1b Study of Trebananib Plus Paclitaxel and Trastuzumab in Patients With HER2-Positive Locally Recurrent or Metastatic Breast Cancer. Clin Breast Cancer. 2019 Feb;19(1):47-57. doi: 10.1016/j.clbc.2018.09.012. Epub 2018 Oct 9. PMID 30420181
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com